CLINICAL TRIAL: NCT04114448
Title: Therapeutic Exercise: Does it Improve Pain Perception, Range of Movement and Quality of Life in Patients With Hemophilia
Brief Title: Therapeutic Exercise in Patients With Hemophilia
Acronym: Hemofisio
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Study was terminated due to lack of funding for continuing
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Alberto Marcos Heredia-Rizo, Assistant Professor. Physiotherapy Department, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HemoFisio2020
Record Dates: First submitted 2019-09-27; First posted 2019-10-03 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-05

CONDITIONS: Hemophilia
Keywords: Hemophilia; Therapeutic exercise; Physical therapy; Randomized controlled trial; Pain perception; Range of movement
MeSH Terms: conditions — Hemophilia A | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercise (Experimental): Patients will be trained to perform a therapeutic exercise intervention protocol. The program will be based on active physical activity including strength, balance an coordination exercises, among others. Each initial contact session will last approximately 1 hour. After baseline, participants will be instructed to undergo at least two sessions per week during 3 consecutive months.
  Interventions: Other: Therapeutic exercise
- Usual care (Active Comparator): Patients will be instructed to perform an usual care physical therapy intervention protocol. Participants in this group will be told to undergo gentle self-performed joint mobilization and stretching exercises. Each initial contact session will last approximately 1 hour. After baseline, participants will be instructed to undergo at least two sessions per week during 3 consecutive months.
  Interventions: Other: Usual physical therapy care

INTERVENTIONS:
Other: Therapeutic exercise — Patients will perform an exercise protocol specifically designed for patients with hemophilia that will include exercises focused on improving range of movement, strength, flexibility, balance and coordination as well as diaphragmatic breathing at the start and at the beginning of each session.
  Arms: Therapeutic exercise
Other: Usual physical therapy care — Patients will undergo usual physical therapy treatment for hemophiliacs, based on affected self and gentle joint mobilization and stretching of muscles involved in the affected joints.
  Arms: Usual care

SUMMARY:
Objectives: To assess the efficacy of performing a therapeutic exercise program, compared with usual care, on pain relief, range of movement and self-perceived quality of life in patients with hemophilia

Design: Quantitative, experimental, longitudinal and prospective study.

Subjects: Male patients between 30 and 45 years old, with hemophilia type A or B and with knee, ankle or elbow arthropathy caused by hemophilia. Participants may be undergoing a pharmacologic treatment with intravenous VIII and/or IX factor

Methods: Participants in the experimental group will an intervention based on therapeutic exercise. One therapist will instruct the patients during two sessions (each lasting approximately 1 hour). Participants will be asked to continue this program at least twice a week. Meanwhile, those in the control group will receive usual physical therapy care, based on a more passive approach, including self-assisted joint mobilization and muscle stretching. Those in the control group will be also instructed to perform the protocol at home, at least twice a week. The intervention protocol in both groups will last three months

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of hemophilia type A or hemophilia type B.
* Knee, elbow or ankle arthropathy caused by hemophilia
* Pharmacological treatment based on using VIII or IX factor concentrates.

Exclusion Criteria:

* Presence of VIII FIX inhibitors.
* Having received anti-inflammatory treatment using Arcoxia (Etoricoxib)
* Having undergone a surgical intervention at the target joint.
* Patients enrolled in other research which implies doing physical exercise.

Ages: 30 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold (PPT) in the evaluated muscles. | Change from baseline to 3 months after intervention
  The PPT levels will be evaluated in KPa. PPT levels, defined as the minimum necessary pressure to evoke pain will be evaluated using a handheld electronic pressure algometer.
Self-reported pain intensity: Numeric Pain Rating Scale (NPRS) | Change from baseline to 3 months after intervention
  Self-reported pain will be evaluated using the Numeric Pain Rating Scale (NPRS), where 0 denotes no pain at all, and 10 denotes the maximum possible pain.
Range of movement (ROM). | Change from baseline to 3 months after intervention
  Active ROM of the affected joint will be evaluated using inertial sensors, that measure lineal acceleration and angular velocity.
General flexibility | Change from baseline to 3 months after intervention
  General flexibility will be assessed using the improved tot-flex test, which makes possible to extrapolate general flexibility from a combined movement measure.
Daily life activities | Change from baseline to 3 months after intervention
  Ordinary daily life activities will be assessed using the Haemophilia Activities List, which measures the self-perceived functional state.
Self-perceived quality of life: A36 Haemophilia-QoL test | Change from baseline to 3 months after intervention
  Quality of life will be evaluated using the A36 Haemophilia-QoL test. This is a valid and specific tool for hemophiliac adults.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto M Heredia-Rizo, PhD, Principal Investigator — Physiotherapy Department, University of Sevilla, Spain
Locations (1):
- University of Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No